CLINICAL TRIAL: NCT00916318
Title: Overweight and Obesity in Preschool Children, Prevalence and Prevention - Family Based Health Interventions for Child Health
Brief Title: Childhood Overweight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vardalinstitutet The Swedish Institute for Health Sciences (Other)
Collaborators: Lund University Hospital (Other)
Responsible Party: Principal investigator: Kristina Thorngren-Jerneck, Lund university Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Obesity-Chrildren Vardal
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-05

CONDITIONS: Childhood Obesity; Childhood Overweight
MeSH Terms: conditions — Pediatric Obesity

ARMS (4):
- A: experimental (Experimental): (A) internet based information and communication tool "Sundabarn.se"(
  Interventions: Behavioral: Obesity-Children
- (B): experimental (Experimental): (B) psychologist directed seminars with different themes, giving parents tools to implement necessary changes in family-patterns and life style, combined with A
  Interventions: Behavioral: Obesity-Children
- (c): experimental (Experimental): (C) occupational therapist directed group-treatment intended to help parents alter their daily life patterns and, combined with A
  Interventions: Behavioral: Obesity-Children
- (D): control group (Active Comparator)
  Interventions: Behavioral: Obesity-Children

INTERVENTIONS:
Behavioral: Obesity-Children — (A) internet based information and communication tool "Sundabarn.se"(B) psychologist directed seminars with different themes, giving parents tools to implement necessary changes in family-patterns and life style, combined with A, (C) occupational therapist directed group-treatment intended to help parents alter their daily life patterns and, combined with A, (D) control group.

SUMMARY:
To evaluate the effects of a family-based intervention program intended for parents of pre-school children (4-6 y) with overweight and obesity (according to Cole et al), and to investigate if treatment has an effect on metabolic parameters. In a randomised controlled trial evaluate the three separate family based intervention programs and to investigate if treatment has an effect by correlating the parameters described above with BMI, before and after the intervention program.

DETAILED DESCRIPTION:
The aim is to investigate the possibility of preventing the development of obesity in early childhood. To evaluate the effects of a family-based intervention program intended for parents of pre-school children (4-6 y) with overweight and obesity (according to Cole et al), and to investigate if treatment has an effect on metabolic parameters. To compare different methods of treatment by randomizing the families into groups with various treatment during one year; (A) internet based information and communication tool "Sundabarn.se"(B) psychologist directed seminars with different themes, giving parents tools to implement necessary changes in family-patterns and life style, combined with A, (C) occupational therapist directed group-treatment intended to help parents alter their daily life patterns and, combined with A, (D) control group. To analyse the aetiology and prognosis of overweight and obesity in early childhood, by measuring the following variables: heredity, genetics, perinatal, physiological, metabolism, bio-chemical, clinical, psychological, socio-economic. In a randomised controlled trial evaluate the three separate family based intervention programs and to investigate if treatment has an effect by correlating the parameters described above with BMI, before and after the intervention program. To calculate the prevalence of overweight and obesity among pre-school children in the county of Middle Skåne during a 20 year period. To analyse parents actual utilization of the Sundabarn.se and in association with primary and secondary outcome. To analyse the cost-effectiveness of the intervention programs.

The primary outcome variable, BMI of the children, is measured at inclusion, after six months, at exclusion and one year after end of program.

Following variables are investigated and related to BMI of children before and after intervention: Heredity: BMI of parents, history . Socio-economic background: education, salary, language, occupation of parents. Perinatal data: Mothers BMI, parity, smoking, ponderal index of infant, gender, breast-feeding. Psychological variables: grading of parents experienced stress and control and psychological health of the child, before end after intervention. Are there a correlation between change in these factors and change in BMI of the child after the intervention? Physiological variables: Sleep duration and activity patterns in the children and compare them to BMI Analysing sleep duration and activity with an accelerometer. Analysing dietary of children: diet registration Analysing the change of bio-chemical markers in blood of children before and after intervention: metabolism of insulin (glc, insulin, C-peptide, pro-insulin, HBA1C) lipids (TG, HDL, LDL, cholesterole), adipokins and cytokins (leptin, adinopektin, resistin, haptoglobulin, IL-6, TNFalfa),ghrelin before and after a meal, thyroid (TSH, T3). Analysing the bacteria of the gastro-intestinal tract by sample from stools.

Utilization of SundaBarn.se: automatic, electronic measurement by single user identity of number of sessions, pages visited, inputs made and downloads.

Intervention health-care resource use: Protocol driven visits to physician, nurse, occupational therapist, psychologist, dietitian.

ELIGIBILITY:
Inclusion Criteria:

* 4-6 y
* BMI due to Cole criteria as overweight or obesity

Exclusion Criteria:

* Medical disorders
* Endocrine disorders

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-12 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: BMI | 6 months, 1 year, 2 year, 5 year

SECONDARY OUTCOMES:
Secondary Outcome Measures: diet registration Analysing the change of bio-chemical markers in blood of children before and after intervention | 6 months, 1 year, 2 year, 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University Childrens' hospital, Lund, Sweden

REFERENCES:
- [Derived] Onnerfalt J, Erlandsson LK, Orban K, Broberg M, Helgason C, Thorngren-Jerneck K. A family-based intervention targeting parents of preschool children with overweight and obesity: conceptual framework and study design of LOOPS- Lund overweight and obesity preschool study. BMC Public Health. 2012 Oct 17;12:879. doi: 10.1186/1471-2458-12-879. PMID 23072247